CLINICAL TRIAL: NCT06418971
Title: Testing & Refinement of CarePair: An Assessment and Referral Platform to Support Family Caregivers of Alzheimer's Disease and Related Dementias.
Acronym: CarePair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Francesca B Falzarano, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UP-25-00690; R00AG073509 (NIH)
Record Dates: First submitted 2024-02-27; First posted 2024-05-17 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Caregiver Burden; Caregiver Burnout; Dementia
Keywords: Dementia family caregivers
MeSH Terms: conditions — Caregiver Burden; Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Participants randomized to the control arm will receive access to an attention-matched comparator: a digital folder containing the same caregiving articles available in the CarePair app. However, the materials will not be personalized or organized. Participants will be asked to log into the digital folder twice per week and read one article at each login, for a total of 12 logins and articles over the 6-week study period, mirroring the engagement frequency of the intervention group.
- CarePair Intervention Arm (Experimental): Participants randomized to the intervention arm will receive access to the CarePair app, a needs-based digital platform that delivers tailored recommendations for Alzheimer's disease and related dementias (ADRD) resources designed for family caregivers. These include services and educational articles personalized based on the caregiver's self-reported needs and preferences, with content organized by relevance to each user. Participants will be asked to log into the CarePair app twice per week and engage with one article per login, for a total of 12 logins and articles over the 6-week study period.
  Interventions: Behavioral: CarePair

INTERVENTIONS:
Behavioral: CarePair — This study will pilot test the feasibility and acceptability of a digital self-assessment and referral tool using machine learning models to enhance service use and address unmet needs in ADRD caregivers.
  Arms: CarePair Intervention Arm

SUMMARY:
The purpose of this study is to develop and test CarePair, a mobile application-based needs assessment and service referral platform for family caregivers of persons with dementia designed to alleviate stress and promote psychosocial well being.

The main aims of this study are:

* To evaluate the feasibility and acceptability of the CarePair mobile application.
* To explore the potential for CarePair to reduce feelings of depression and burden, and improve caregivers' feelings of self-efficacy.

Caregiver participants will be asked to log in and use the CarePair application and complete study activities for a six-week duration. Researchers will compare the intervention group to an attention control comparator to see if application use is associated with improved psychosocial outcomes at follow-up.

DETAILED DESCRIPTION:
In 2024, approximately 6.9 million diagnosed cases of Alzheimer's disease and related dementias (ADRD) were reported in the United States, with 83% of the caregiving burden shouldered by unpaid family members or friends. The duration of ADRD varies between 4-20 years, during which individuals often transition into a state of complete dependency. Without family caregivers, the long-term services and support system would be unsustainable. The dearth of accessible support for ADRD caregivers constitutes a significant public health emergency. Caregivers are frequently uncertain of which services are needed, available, and how to gain access - often leaving those most vulnerable without essential support. When queried about service underuse, study respondents who participated in the K99 phase of this project highlighted an information deficit tailored to specific cultures, demographics, and dementia types. They described the excess of online information as overwhelming, often irrelevant, impractical, or unaffordable. Existing technology-based solutions targeted toward enhancing personalized caregiver support are limited. Leveraging continued innovations in technology to inform the training and testing of machine learning algorithms, which can match and update resources while accounting for individual needs, preferences (in-person, virtual), and barriers (e.g., employment, lack of respite care), holds great potential to enhance the precision of service linkage for ADRD caregivers. This R00 project aims to develop, refine, and pilot test CarePair (formerly the Caregiver Resource Room), a mobile application assessment and service referral platform for dementia caregivers. CarePair will leverage innovative machine learning algorithms to holistically evaluate caregivers' evolving needs, their barriers, and preferences to generate personalized service referrals relevant to their areas of identified need. Thus, the specific aims of the R00 are to 1) Use mixed-method and focus group data from the K99 phase to inform the iterative development of the CarePair, which includes a digital self-assessment tool employing machine learning to identify needs, categorize them, and generate targeted service recommendations; 2) Evaluate front- and back-end usability (e.g., via task analysis, heuristic evaluation) of the tool's content, design, features, functionality, and accuracy of service output. Feedback will inform modifications and iterative refinement of the CarePair Version 2.0; 3) Conduct a pilot randomized controlled trial to assess the feasibility, acceptability, and preliminary efficacy of CarePair in enhancing service awareness, addressing unmet needs, and improving mental health. The proposed research aligns with the NIA's strategic initiative to foster research scientists in aging and to develop promising interventions to better engage and support the well-being of ADRD family caregivers.

ELIGIBILITY:
Inclusion:

* Currently a primary caregiver of a community-dwelling PwD
* Provides at least 10 hours of care per week
* ≥18 years of age
* Fluent in English
* Both the caregiver and care-recipient reside in and/or can easily access one of the following cities/areas: New York City, New York (NY); Long Island, NY; Westchester County, NY; Seattle, Washington (WA); Los Angeles, California (CA)
* Provides at least 10 hours of care per week
* Has provided care for at least 6 months
* Able to use the internet and has internet access
* Owns and can operate a smartphone
* Able and willing to provide their informed consent to participate for the six-week study duration
* Does not self-report any cognitive impairments

Exclusion:

* Not currently the primary caregiver of a community-dwelling person with dementia
* Care-recipient lives in residential care (e.g., assisted living, skilled nursing facility)
* ≤18 years of age
* Not fluent in English
* The caregiver and/or care-recipient resides outside of and/or cannot easily access any of the following cities: New York City (NY); Long Island (NY); Westchester County (NY); Seattle (WA); Los Angeles (CA)
* Provides less than 10 hours of care per week
* Has provided care for less than 6 months
* Unable to use the internet or does not have internet access
* Does not own and/or cannot operate a smartphone
* Unable or unwilling to provide informed consent to participate for the six-week study duration
* Self-reports having a cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The Feasibility of the CarePair study as measured by the proportion of family caregivers who complete the study screening survey. | Enrollment
  The feasibility of the CarePair study will be measured by the proportion of family caregivers who complete the study screening survey among those who were directly invited to participate the study.
The Feasibility of the CarePair study as measured by the proportion of family caregivers who consent to participate and are enrolled. | Enrollment
  The feasibility of the CarePair study will be measured by the proportion of family caregivers who consent to participate among those who were screened into the study. Participants who consent to participate are then immediately randomized to their assigned condition and thus enrolled.
The Feasibility of the CarePair study as measured by the proportion of are deemed eligible based on screening criteria. | Enrollment
  The feasibility of the CarePair study will be measured by the proportion of family caregivers who are deemed eligible to participate based on screening criteria among those who completed the study's screening survey.
The Feasibility of the CarePair study as measured by recruitment rates and the proportion of family caregivers that decline participation. | Enrollment
  The feasibility of the CarePair study will be measured by the proportion of eligible family caregivers who decline to participate among those who were screened into the study.
The Feasibility of the CarePair study as measured by participant retention, as indicated by the number of participants lost to follow-up. | Enrollment to 6-Week Follow-Up
  Participant retention, as an aspect of feasibility, will be measured by the recorded number of participants number lost to follow-up. A number of the enrolled participants who the study team contacted weekly for 4 weeks, but did not answer or continue participation, will be recorded.
The Feasibility of the CarePair study as measured by participant retention, as indicated by the number of recorded dropouts. | Enrollment to 6-Week Follow-Up
  Participant retention, as an indicator of feasibility, will be assessed by recording the number of participants who withdraw from the study after enrollment
The Feasibility of the CarePair application as measured by the number of app logins per participant out of total required (minimum= 12). | Baseline to 6-Week Follow-Up
  The feasibility of the application will be measured by the number of times the participant logs in to the CarePair application. The minimum number of logins recommended to the participants is 12 (2x/week for 6 weeks).
The Feasibility of the CarePair application as measured by the number of app interactions per participant out of total required (minimum= 12). | Baseline to 6-Week Follow-Up
  Feasibility of the application will be assessed based on the number of participant interactions with CarePair's features, such as reviewing, rating, taking notes on, or saving services or articles. Participants are asked to log in and engage with the app approximately twice per week over the six-week study period, for a recommended minimum of 12 total interactions.
Application Usability, as measured using the validated System Usability Scale (SUS). | 6-Week Follow-Up
  Usability and accessibility of the CarePair application design will be measured using the validated System Usability Scale (SUS). Total scores for the SUS range from 0-100, with higher scores indicative of greater usability. A threshold score of 68 is used to indicate adequate usability.
Application usability, as measured using the validated User Version of the Mobile App Rating Scale (uMARS). | 6-Week Follow-Up
  Usability of the CarePair application will be measured using the validated user version of the Mobile App Rating Scale (uMARS). The uMARS provides a multidimensional assessment of app quality, including engagement, functionality, aesthetics, and information. Scores range from 20 to 100, with higher scores indicating more favorable user evaluations of the app's usability and overall quality.
The Acceptability of the CarePair application as measured by a survey that measures the participants satisfaction and acceptability of the application. | 6-Week Follow-Up
  The acceptability of the CarePair application will be measured by the use of surveys assessing usability, engagement, acceptability, suggestions for improvement.
  Participants will be asked to rate their agreement with statements including "I enjoyed my experience using the CarePair application". Response options are rated on a five-point scale from 1-Strongly Disagree to 5-Strongly Agree. Scores range from 9-45, with higher scores indicating greater satisfaction and acceptability.
The Acceptability of the CarePair application as measured by a qualitative survey that measures the participants satisfaction and acceptability of the application. | 6-Week Follow-Up
  The acceptability of the CarePair application will be measured by the use of open-ended items assessing usability, engagement, acceptability, suggestions for improvement. The intervention group participants will be administered five open-ended qualitative items asking for feedback on CarePair. Sample items include: "Would you continue using the CarePair application after this study? Why or why not?"

SECONDARY OUTCOMES:
Change from Baseline Caregiver Needs scores on a 12-item Needs Assessment | Baseline; 6-Week Follow-Up
  A 12-item caregiver needs assessment will be used to measure family caregivers' care-related needs, such as legal guidance, social support, and education. Total scores range from 12-48, with higher scores representing greater caregiver needs.
Change from Baseline Caregiving Self-Efficacy scores on the 15-item Revised Scale for Caregiving Self-Efficacy | Baseline; 6-Week Follow-Up
  Caregiving Self-Efficacy will be measured using the Revised Scale for Caregiving Self-Efficacy. Total scores range from 0-100, with higher scores indicative of greater feelings of perceived self-efficacy.
Change from Baseline Caregiver Depressive Symptoms as measured by the Patient Health Questionnaire-9 (PHQ-9). | Baseline; 6-Week Follow-Up
  The PHQ-9 will be used to measure family caregiver depressive symptoms. Total scores range from 0-27, with higher scores indicative of greater caregiver depressive symptoms.
Change from Baseline Anxiety scores on the Generalized Anxiety Disorder-7 (GAD-7) | Baseline; 6-Week Follow-Up
  Change in caregivers' anxiety scores will be assessed using the GAD-7. Scores range from 0-21, with higher scores indicating a greater level of anxiety.
Change from Baseline Caregiver Stress as measured by the Kingston Caregiver Stress Scale (KCSS) | Baseline; 6-Week Follow-Up
  The KCSS will be used to measure family caregiver stress. Total scores range from 20-50, with higher scores indicative of greater caregiver stress.
Change from Baseline Quality of Life scores on the 5-item Satisfaction with Life Scale (SWLS) | Baseline; 6-Week Follow-Up
  The SWLS will be used to measure family caregiver quality of life. Total scores range from 5-35, with a score of 20 representing a neutral point on the scale. Higher scores indicate a greater level of satisfaction with life.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Falzarano, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected for the CarePair study will only be shared after the investigators have published the data addressing the study's specific aims. Intellectual property and data generated under this project will be administered in accordance with both University of Southern California (USC) and NIH policies, including the NIH Data Sharing Policy and Implementation Guidance. After publication of the investigator's main findings, access to databases and associated software tools generated and the code to create these tools under the project will be available for educational, research and non-profit purposes.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: These data will be shared after the investigators have published the specific aims of this study. Requests for the code used to create CarePair will be reviewed by the investigative team and shared once feasibility, acceptability, and preliminary efficacy has been examined and the findings have been published.
Access Criteria: Individuals who wish to access the data are required to: 1) Use the data for research purposes only; 2) Not identify any individual participant; 3) Secure the data using appropriate computer technology such as password-protected servers and files; and 4) Return and/or destroy data after analyses are complete.